CLINICAL TRIAL: NCT01563640
Title: Can Insecticide-treated School Uniforms Reduce Dengue Infections in School-aged Children in Thailand
Brief Title: Insecticidal School Uniforms for Dengue Prevention in Thailand
Acronym: DengueTools
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Insecticidal treatment of school uniforms did not last through a dengue season
Sponsor: Umeå University (Other)
Collaborators: European Union (Other)
Responsible Party: Principal Investigator, Peter Byass, Professor of Global Health, Umeå University
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 282589-T
Record Dates: First submitted 2012-03-16; First posted 2012-03-27 (Estimated); Last update posted 2015-09-01 (Estimated); Status verified 2015-08

CONDITIONS: Dengue
Keywords: dengue
MeSH Terms: conditions — Dengue | interventions — Therapeutic Irrigation

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- normal school uniforms (Placebo Comparator): washing only
  Interventions: Other: washing
- insecticide-treated school uniforms (Experimental): washing and insecticide treatment
  Interventions: Other: permethrin insecticide

INTERVENTIONS:
Other: permethrin insecticide — commercial permethrin insecticide impregnation of clothing before transmission season
  Arms: insecticide-treated school uniforms
Other: washing — normal washing of school uniforms, without permethrin insecticide impregnation
  Arms: normal school uniforms

SUMMARY:
This is a randomised controlled trial that will be conducted in eastern Thailand in a group of schools with approximately 2,000 students aged 7-15 years. Pre-fabricated school uniforms will be commercially treated to ensure consistent high quality of insecticide impregnation with permethrin. A double-blind randomised cross-over trial at the school level will cover two dengue transmission seasons.

ELIGIBILITY:
Inclusion Criteria:

* pupils in participating schools

Exclusion Criteria:

* skin sensitivity, exema

Ages: 7 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1825 (Actual)
Dates: Start 2012-03; Primary Completion 2013-06 (Actual); Study Completion 2014-12 (Actual)

PRIMARY OUTCOMES:
insecticide:placebo incidence rate-ratio (per 1,000 person-years) of laboratory-confirmed dengue cases in school-aged children | up to 2 years
  Schools are cross-over randomised to insecticide-treated or untreated (placebo) school uniforms, and so the primary outcome is the rate-ratio of dengue fever cases in school children, compared between these two groups.

SECONDARY OUTCOMES:
comparison between intervention and placebo groups of number of serious skin reactions to insecticide-treated uniforms | up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Annelies Wilder-Smith, MD, Principal Investigator — Umeå University
Locations (1):
- Centre of Excellence for Vectors and Vector-Borne Diseases, Mahidol University, Salaya, Thailand

REFERENCES:
- [Derived] Kittayapong P, Olanratmanee P, Maskhao P, Byass P, Logan J, Tozan Y, Louis V, Gubler DJ, Wilder-Smith A. Mitigating Diseases Transmitted by Aedes Mosquitoes: A Cluster-Randomised Trial of Permethrin-Impregnated School Uniforms. PLoS Negl Trop Dis. 2017 Jan 19;11(1):e0005197. doi: 10.1371/journal.pntd.0005197. eCollection 2017 Jan. PMID 28103255
- [Derived] Wilder-Smith A, Byass P, Olanratmanee P, Maskhao P, Sringernyuang L, Logan JG, Lindsay SW, Banks S, Gubler D, Louis VR, Tozan Y, Kittayapong P. The impact of insecticide-treated school uniforms on dengue infections in school-aged children: study protocol for a randomised controlled trial in Thailand. Trials. 2012 Nov 15;13:212. doi: 10.1186/1745-6215-13-212. PMID 23153360
- See also: Related Info — http://www.denguetools.net